CLINICAL TRIAL: NCT01221129
Title: Zinc and the Synthesis of Zinc Binding Proteins (Protocol B)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: UF-GCRC-772; R01DK031127 (NIH)
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Zinc Deficiency
Keywords: zinc; reticulocyte; PBMC; whole blood; transcriptome; microarray
MeSH Terms: interventions — Acclimatization; Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic; Clinical Trials, Phase III as Topic

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood cells in clotted blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dietary Restriction
  Interventions: Other: Acclimation; Other: Dietary zinc depletion; Other: Dietary zinc repletion

INTERVENTIONS:
Other: Acclimation — 11 mg Zn/day as a controlled intake level
  Other Names: Adaptation; Phase 1
Other: Dietary zinc depletion — < 1 mg Zn/day achieved by providing a liquified diet of defined nutrient content
  Other Names: Phase 2
Other: Dietary zinc repletion — 15 mg Zn/day as a daily supplement plus normal habitual diet without restriction
  Other Names: Phase 3

SUMMARY:
The specific aim of this protocol is to examine differential expression of specific mRNAs and proteins that occur when the dietary intake of zinc is acutely reduced below the dietary requirement for a period of ten days.

DETAILED DESCRIPTION:
Methods to assess the dietary zinc status of individual humans or populations are lacking. The study is a three period observational study of biomarkers of zinc status before, during and after zinc depletion. The entire dietary study will take 24 days composed of three parts:

* Dietary Acclimation (Phase 1): 7 days
* Dietary Zinc Restriction (Phase 2): 10 days
* Dietary Zinc Repletion (Phase 3): 7 days

The dietary treatments and all blood draws will be carried out in the General Clinical Research Center (GCRC) at University of Florida. Previous research from has shown that both metallothionein gene expression and specific zinc transporter genes in blood leukocyte subsets are directly proportional to dietary zinc intake. By using cDNA array analysis and quantitative PCR technology with blood RNA, those genes most sensitive to zinc nutrition will be identified for the purpose of developing zinc status assessment methods on how zinc functions in human biology.

Additionally, buccal mucosal cells will be collected in the GCRC by using swabs, i.e., in a noninvasive manner, to further characterize the expression pattern of the genes under study. This method has the potential for nutrition studies in the field (international nutrition, etc).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* 21-35 years
* Body weight above 110 lb

Exclusion Criteria:

* Use of dietary supplements
* Smoker
* Alcoholic
* Under medication
* History of chronic disease
* Use of denture cream
* Vegetarian
* Food allergy

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: UF campus community
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Serum zinc concentration | 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Cousins, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Ryu MS, Guthrie GJ, Maki AB, Aydemir TB, Cousins RJ. Proteomic analysis shows the upregulation of erythrocyte dematin in zinc-restricted human subjects. Am J Clin Nutr. 2012 May;95(5):1096-102. doi: 10.3945/ajcn.111.032862. Epub 2012 Mar 28. PMID 22456662